CLINICAL TRIAL: NCT04933201
Title: Music for Postoperative Pain and Discomfort After Orbital Decompression
Brief Title: Postoperative Music for Orbital Decompression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huijing Ye, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202105
Record Dates: First submitted 2021-06-14; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Surgery; Pain; Musth
Keywords: postoperative pain; postoperative discomfort; general anesthesia
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music group (Experimental): Perioperative music intervention
  Interventions: Other: Music
- Control group (Active Comparator): No perioperative music
  Interventions: Other: Routine perioperative treatment

INTERVENTIONS:
Other: Music — Perioperative musical intervention
  Arms: Music group
Other: Routine perioperative treatment — Routine perioperative treatment
  Other Names: Routine perioperative treatment without music
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the effect of music to the postoperative pain and discomfort after orbital decompression.

DETAILED DESCRIPTION:
To investigate the effect of music to the postoperative pain and discomfort after orbital decompression under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 16-75 years old
* diagnosed as thyroid eye disease
* bone removal orbital decompression under general anesthesia

Exclusion Criteria:

* any uncontrolled clinical problems
* orbital decompression under local anesthesia
* Reluctance to participate in clinical trials

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain after orbital decompression | 24 hour after recovery
  Pain levels measured using Numerical Rating Scale (NRS) ranging from 0 to 10, where 0 represents no pain and 10 represents the worst pain imaginable ; this scale has been confirmed to be sensitive and reliable.Clinically significant postoperative pain was considered serious pain (NRS score ≥5).

SECONDARY OUTCOMES:
Discomfort after orbital decompression | 24 hour after recovery
  Discomfort levels were measured using Numerical Rating Scale (NRS) ranging from 0 to 10, where 0 represents no discomfort and 10 represents the worst discomfort; this scale has been confirmed to be sensitive and reliable. Discomfort was defined as "sensation other than pain" and included nausea, vomiting, headache, and dizziness. Clinically significant postoperative discomfort was considered serious discomfort (NRS score ≥5) any time postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Huijing Ye, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided